CLINICAL TRIAL: NCT00080782
Title: A Randomized Phase II Trial of Bone-Targeted Therapy Consisting of Strontium-89 and Doxorubicin With or Without Celecoxib in Androgen-Independent Prostate Cancer
Brief Title: Doxorubicin and Strontium-89 With or Without Celecoxib in Treating Patients With Progressive Androgen-Independent Prostate Cancer and Bone Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual due to competing trial.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-035; P50CA090270 (NIH); P30CA016672 (NIH); MDA-ID-02035 (Other: UT MD Anderson Cancer Center); CDR0000355360 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; bone metastases; Progressive Androgen-Independent Prostate Cancer; Metastron; Sr-89; Strontium-89; strontium chloride Sr 89; Celecoxib; Celebrex; Doxorubicin; Rubex; Adriamycin
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Celecoxib; Doxorubicin; strontium chloride; Strontium-89

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Celecoxib (Experimental): Doxorubicin IV over 30 minutes on days 1, 8, 15, and 22 + Strontium chloride Sr 89 IV on day 1, and oral celecoxib twice daily in absence of disease progression.
  Interventions: Drug: Celecoxib; Drug: Doxorubicin Hydrochloride; Radiation: Strontium chloride Sr 89
- Arm II: No Celecoxib (Experimental): Doxorubicin IV over 30 minutes on days 1, 8, 15, and 22 + Strontium chloride Sr 89 IV on day 1.
  Interventions: Drug: Doxorubicin Hydrochloride; Radiation: Strontium chloride Sr 89

INTERVENTIONS:
Drug: Celecoxib — Oral celecoxib twice daily in the absence of disease progression.
  Other Names: Celebrex
  Arms: Arm I: Celecoxib
Drug: Doxorubicin Hydrochloride — By vein (IV) over 30 minutes on days 1, 8, 15, and 22
  Other Names: Adriamycin; Rubex
Radiation: Strontium chloride Sr 89 — IV on day 1
  Other Names: Sr-89; Metastron; Strontium-89

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Strontium-89 may relieve bone pain caused by prostate cancer. Celecoxib may stop the growth of cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for tumor cell growth. Combining doxorubicin and strontium-89 with celecoxib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying celecoxib together with doxorubicin and strontium-89 to see how well they work compared to doxorubicin and strontium-89 alone in treating patients with progressive androgen-independent prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare time to prostate-specific antigen progression in patients with progressive androgen-independent prostate cancer and bone metastases treated with doxorubicin and strontium chloride Sr 89 with or without celecoxib.

OUTLINE: This is a randomized study. Patients are stratified according to extent of bone metastases on bone scan (> 20 lesions vs ≤ 20 lesions) and quality of response (i.e., decline of the prostate-specific antigen from baseline) to prior induction chemotherapy (≥ 80% vs < 80%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin IV over 30 minutes on days 1, 8, 15, and 22 and strontium chloride Sr 89 IV on day 1. Patients also receive oral celecoxib twice daily in the absence of disease progression.
* Arm II: Patients receive doxorubicin and strontium chloride Sr 89 as in arm I.

PROJECTED ACCRUAL: A total of 70 patients (35 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of androgen-independent prostate cancer

  * Osteoblastic metastases
  * No predominant visceral metastases
* Progressive disease after response to prior induction chemotherapy (prostate-specific antigen decline of at least 50% from baseline after 16 weeks of treatment)
* No symptomatic lymphadenopathy (i.e., scrotal or pedal edema)

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Adequate physiologic reserves

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* No prior radionuclide therapy

Surgery

* Not specified

Other

* No more than 3 prior cytotoxic treatments
* More than 6 months since prior celecoxib or rofecoxib

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-02; Primary Completion 2004-04 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Time to prostate-specific antigen progression | Continuous assessment 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Tu, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org